CLINICAL TRIAL: NCT02017821
Title: The Effect of Aerobic Endurance Training in Patients With Drug Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/639
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Substance-Related Disorders
Keywords: Exercise; Oxygen Consumption; mental health
MeSH Terms: conditions — Substance-Related Disorders; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- training group (Experimental): high intensity aerobic training 3 weekly sessions for 8 weeks
  Interventions: Behavioral: high intensity aerobic training
- care as usual (No Intervention)

INTERVENTIONS:
Behavioral: high intensity aerobic training
  Arms: training group

SUMMARY:
Physical health does not have a high priority in today's treatment of patients with substance use disorder (SUD) patients have a poor physical health not only due to injuries related to the substance abuse, but also because of the lifestyle that addiction causes. There are today few studies that provide information about SUD patients' physical health. One of the project's aims is to document the physical health of SUD patients in treatment, using objective measures. After completion of various physical tests, an 8 week period of high intensity aerobic training intervention will follow. It will be investigated if the SUD patients are able to engage and participate throughout the whole training intervention, to what degree the participants improve their physical health and the effect of physical health improvement on substance abuse treatment.

ELIGIBILITY:
Inclusion Criteria:

* substance use disorder diagnosed ICD10
* written informed consent
* "residential treatment"

Exclusion Criteria:

* not been using drugs the last six months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-08; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
change in maximal oxygen consumption (VO2 max) | from baseline to 8 weeks
  Directly measurement of maximal oxygen consumption. Measurement of work efficiency and lactate measurements. Insomnia Severity Index and Hospital Anxiety and Depression scale is used to measure mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Eivind Wang, phd, Study Director — Norwegian University of Science and Technology
Locations (1):
- Trondheims Klinikken, St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Flemmen G, Unhjem R, Wang E. High-intensity interval training in patients with substance use disorder. Biomed Res Int. 2014;2014:616935. doi: 10.1155/2014/616935. Epub 2014 Mar 2. PMID 24724089